CLINICAL TRIAL: NCT06230471
Title: A Phase II, Multicenter, Randomized Study of Pembrolizumab With or Without Chemotherapy or Lenvatinib in First-Line Treatment of Advanced Biliary Tract Cancer
Brief Title: Pembrolizumab With or Without Lenvatinib or Chemotherapy in First-Line Treatment of Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K5033
Record Dates: First submitted 2024-01-10; First posted 2024-01-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Neoplasms Immunotherapy
MeSH Terms: interventions — pembrolizumab; lenvatinib; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab,Lenvatinib and Gemox Chemotherapy（Gemcitabine and Oxaliplatin） (Experimental): Drug：Pembrolizumab Pembrolizumab 200 mg will be administered intravenously once every three weeks, with intravenous infusion on Day 1 of each cycle. Drug: Lenvatinib Oral Product The dose of lenvatinib is 12mg/day for patients with a body weight of ≥60 kg, and 8mg/day for patients with a body weight of <60 kg, taken once daily. Drug: Chemotherapy GEMOX regimen: Gemcitabine 1000mg/m2 will be administered intravenously over 30 minutes on Day 1 and Day 8; Oxaliplatin 100mg/m2 will be administered intravenously over 2 hours on Day 1, and the cycle will be repeated every 3 weeks
  Interventions: Drug: Pembrolizumab,Lenvatinib and Gemox Chemotherapy（Gemcitabine and Oxaliplatin）
- Pembrolizumab and Lenvatinib (Experimental): Drug：Pembrolizumab Pembrolizumab 200 mg will be administered intravenously once every three weeks, with intravenous infusion on Day 1 of each cycle. Drug: Lenvatinib Oral Product The dose of lenvatinib is 12mg/day for patients with a body weight of ≥60 kg, and 8mg/day for patients with a body weight of <60 kg, taken once daily.
  Interventions: Drug: Pembrolizumab and Lenvatinib
- Pembrolizumab and Gemox Chemotherapy（Gemcitabine and Oxaliplatin） (Active Comparator): Drug：Pembrolizumab Pembrolizumab 200 mg will be administered intravenously once every three weeks, with intravenous infusion on Day 1 of each cycle. Drug: GEMOX Chemotherapy GEMOX regimen: Gemcitabine 1000mg/m2 will be administered intravenously over 30 minutes on Day 1 and Day 8; Oxaliplatin 100mg/m2 will be administered intravenously over 2 hours on Day 1, and the cycle will be repeated every 3 weeks
  Interventions: Drug: Pembrolizumab and Gemox Chemotherapy（Gemcitabine and Oxaliplatin）

INTERVENTIONS:
Drug: Pembrolizumab,Lenvatinib and Gemox Chemotherapy（Gemcitabine and Oxaliplatin） — Drug: Pembrolizumab Pembrolizumab 200 mg will be administered intravenously once every three weeks, with intravenous infusion on Day 1 of each cycle. Drug: Lenvatinib Oral Product The dose of lenvatinib is 12mg/day for patients with a body weight of ≥60 kg, and 8mg/day for patients with a body weight of <60 kg, taken once daily. Drug: Chemotherapy GEMOX regimen: Gemcitabine 1000mg/m2 will be administered intravenously over 30 minutes on Day 1 and Day 8; Oxaliplatin 100mg/m2 will be administered intravenously over 2 hours on Day 1, and the cycle will be repeated every 3 weeks.
  Arms: Pembrolizumab,Lenvatinib and Gemox Chemotherapy（Gemcitabine and Oxaliplatin）
Drug: Pembrolizumab and Lenvatinib — Pembrolizumab and Lenvatinib
  Arms: Pembrolizumab and Lenvatinib
Drug: Pembrolizumab and Gemox Chemotherapy（Gemcitabine and Oxaliplatin） — Pembrolizumab and Gemox Chemotherapy（Gemcitabine and Oxaliplatin）
  Arms: Pembrolizumab and Gemox Chemotherapy（Gemcitabine and Oxaliplatin）

SUMMARY:
Explore the impact of the first-line application of Pembrolizumab with or without Lenvatinib or chemotherapy, on the survival, disease progression, and drug safety of patients with advanced biliary tract cancers

DETAILED DESCRIPTION:
This trial is a three-arm, randomized, multi-center clinical study. Eligible subjects who meet the study criteria will be screened and randomized in a 1:1:1 ratio to receive treatment with intravenous infusion of Pembrolizumab with or without chemotherapy and oral lenvatinib. The investigators will closely follow up and assess the efficacy and safety of the combined treatment, evaluate the progression-free survival of the subjects until progression occurs, and observe their overall survival as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* • The subjects voluntarily participate in the study and agree to sign the informed consent form, are compliant, and cooperate with follow-up.

  * They are over 18 years of age and gender is not restricted when signing the informed consent form.
  * They have histologically confirmed unresectable advanced or metastatic biliary tract adenocarcinoma, including intrahepatic or extrahepatic cholangiocarcinoma and gallbladder cancer.
  * Patients who are diagnosed with unresectable or metastatic disease and have not received prior treatment are eligible for inclusion.
  * Patients who have undergone curative surgery and experienced disease recurrence after more than 6 months; or patients who have completed adjuvant therapy (chemotherapy and/or radiotherapy) and have been disease-free for more than 6 months after completing adjuvant therapy are eligible for inclusion.
  * They have at least one measurable lesion (as defined by RECIST 1.1, the measurable lesion is a spiral CT scan long diameter ≥10mm or lymph node short diameter ≥15mm).
  * Their ECOG score is 0-1 in the week prior to enrollment.
  * Based on the investigator's assessment, their estimated survival time is ≥3 months.
  * Patients with active hepatitis B or C require relevant antiviral treatment, with HBV-DNA <2000 IU/ml (<104 copies/ml), and have received at least 14 days of antiviral treatment before participating in the study. HCV RNA-positive patients must follow local standard treatment guidelines for antiviral therapy, and their liver function is within CTCAE Grade 1 elevation.
  * Their hematological and organ functions are adequate, based on laboratory test results obtained within 14 days before the start of the study (unless otherwise specified):
  * Hematology: (no blood transfusion, no G-CSF, no drug correction within 14 days prior to screening) Hb ≥90 g/L; neutrophil count ≥1.5×109/L; PLT

    ≥100×109/L.
  * Biochemistry: (no albumin transfusion within 14 days) Appropriate liver function: ALT and AST ≤2.5×ULN; for patients with liver metastases, ALT and AST ≤5 × ULN. Serum bilirubin ≤2.0×ULN; these conditions do not apply to patients with confirmed Gilbert's syndrome. Any clinically significant biliary obstruction should be resolved before randomization. Appropriate renal function: creatinine ≤1.5×ULN, or creatinine clearance rate (CCr) >50mL/min (using the standard Cockcroft-Gault formula): Female: CrCl = ((140 - age) x weight (kg) x 0.85) / 72 x serum creatinine (mg/ dL) Male: CrCl = ((140 - age) x weight (kg) x 1.00) / 72 x serum creatinine (mg/ dL)

    * Women of childbearing potential: agree to abstain from sexual intercourse or use contraceptive methods with a failure rate of less than 1% during the treatment period and for at least 6 months after the last dose. If a female patient has menstruation and has not reached menopause (continuous absence of menstruation for ≥12 months without other reasons), and has not undergone sterilization surgery (removal of ovaries and/or uterus), she is considered to be of childbearing potential. Examples of contraceptive methods with a failure rate of less than 1% include bilateral tubal ligation, male sterilization, hormone-based contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual restraint should be evaluated relative to the duration of the clinical trial and the patient's preferred lifestyle and daily routine. Periodic abstinence (such as calendar day, ovulation period, symptom temperature, or post-ovulation method) and ejaculation outside the vagina are unacceptable contraceptive methods.
    * Male: agree to abstain from sexual intercourse or use contraceptive measures, agree not to donate sperm, as defined below: When the female partner is of childbearing potential, male patients must abstain during the treatment period and for 6 months after the last dose, or use a condom plus other contraceptive methods to achieve a failure rate of less than 1%. Male patients must also agree not to donate sperm during the same period. When the female partner is already pregnant, male patients must abstain or use a condom to prevent fetal exposure to the study during the treatment period and for 6 months after the last dose. The reliability of sexual restraint should be evaluated relative to the duration of the clinical trial and the patient's preferred lifestyle and daily routine. Periodic abstinence (such as calendar day, ovulation period, symptom temperature, or post-ovulation method) and ejaculation outside the vagina are unacceptable contraceptive methods.

Exclusion Criteria:

* • Previous systemic treatment received.

  * ECOG score > 1.
  * Pancreatic cancer.
  * Pregnant (positive pregnancy test before medication) or breastfeeding women.
  * Known allergy or intolerance to recombinant humanized PD-1 monoclonal antibody drugs, lenvatinib and its components (or any excipients).
  * Received local anti-tumor treatment within 4 weeks before the first study drug treatment, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection (allowing palliative radiotherapy for bone metastases at least 2 weeks before study drug treatment).
  * Previous or existing grade 3 or higher gastrointestinal fistula or non gastrointestinal fistula (such as skin) according to CTCAE 5.0 criteria.

Multiple factors affecting oral administration of lenvatinib (such as inability to swallow, chronic diarrhea and intestinal obstruction, or other conditions that significantly affect drug intake and absorption).

* Major surgery (except biopsy) has been performed within 4 weeks before the first study drug treatment, or the surgical incision has not completely healed; minor surgery (such as simple excision, biopsy, etc.) was performed within 7 days before the first study intervention.
* Significant cardiovascular and cerebrovascular diseases, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, cerebrovascular accidents or transient ischemic attacks within 6 months before enrollment, congestive heart failure (New York Heart Association classification ≥2), arrhythmia requiring antiarrhythmic drugs (except beta blockers or digoxin), and repeated electrocardiogram showing QTc interval >480 milliseconds (ms). Hepatic or renal dysfunction, with manifestations such as jaundice, ascites, and/ or bilirubin >3×ULN, creatinine ratio >3.5g/24 hours, or renal failure requiring blood or peritoneal dialysis, and/or urinary routine showing urine protein ≥++ or confirmed 24-hour urine protein quantification >1.0g.
* Persistent infection > grade 2 (CTCAE 5.0).
* History of thrombotic events (including stroke and/or transient ischemic attacks) within the past 6 months.
* Poorly controlled hypertension (systolic blood pressure >160mmHg, diastolic blood pressure >100mmHg) despite treatment with antihypertensive medications. Active autoimmune disease or history of autoimmune disease within the past 2 years; participants with active, known, or suspected autoimmune diseases that may affect important organ function or require systemic immunosuppressive therapy are excluded, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid syndrome associated with thrombosis, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. However, participants with type 1 diabetes, hypothyroidism requiring only hormone replacement, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or alopecia) or participants who will not relapse without external triggering factors are allowed.

Replacement therapy (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.

* Known active central nervous system (CNS) metastasis and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate as long as they are stable (evidence of no progression on imaging at least 4 weeks before the first trial treatment and any neurological symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not used steroids for at least 7 days before trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability. Participants with known or untreated brain metastases or epilepsy requiring medication are also excluded. Planned or prior organ or allogeneic bone marrow transplantation. Known history of active tuberculosis (Mycobacterium tuberculosis). History of gastrointestinal bleeding within the past 6 months or clear evidence of gastrointestinal bleeding tendencies, such as bleeding esophageal varices, locally active gastrointestinal ulcerative lesions, fecal occult blood ≥(++), cannot be included; if fecal occult blood (+), gastroscopy is required; evidence or history of bleeding mechanism disorders of grade ≥3 (CTCAE 5.0), or other bleeding disorders.

  * Known human immunodeficiency virus (HIV) infection.
  * Known active hepatitis B or C infection and not receiving regular treatment.
  * During the screening period, HBV DNA ≥2000 IU/ml (or ≥104 copies/ ml) must be reduced to <2000 IU/ml (or <104 copies/ml) with entecavir before enrollment. For eligible participants with Anti-HBc (+)/HBsAg (+)/ HBV DNA< 2000 IU/ml or Anti-HBc (+)/HBsAg (-)/HBV DNA< 2000 IU/ ml, antiviral therapy must be administered during the trial period using the original medication or entecavir or tenofovir.
  * Severe non-healing wounds, ulcers, or fractures.
  * History of substance abuse or any medical, psychological, or social condition that may affect the study, patient compliance, or endanger patient safety.
  * Unresolved toxicity of grade >1 (CTCAE 5.0) caused by any prior treatment/procedure, except for hair loss, anemia, and hypothyroidism.
  * Severe non-healing wounds, ulcers, or fractures.
  * Objective evidence of severe pulmonary impairment, such as a history of severe pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, or drug-related pneumonia.
  * Treatment with a strong CYP3A4 inhibitor (e.g., clarithromycin, indinavir, itraconazole, lopinavir, nelfinavir, ritonavir, saquinavir, telaprevir, voriconazole, etc.) within 7 days before participating in the study, or treatment with a strong CYP3A4 inducer (e.g., phenytoin, phenobarbital, primidone, carbamazepine, rifampin, rifabutin, rifapentine, or St. John's Wort) within 12 days before participating in the study.
  * Concomitant malignancy, except for previously treated skin basal cell carcinoma, squamous cell carcinoma, carcinoma in situ of the breast or cervix, superficial bladder cancer that has been treated, and prostate cancer that has been treated with surgery and has a normal range of PSA tumor markers, or any other malignancy that has not been cured within the past 5 years.
  * The investigator determines that the participant is unsuitable for the study based on overall medical condition.
  * Concurrent participation in another clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Baseline up to approximately 6 months
  Objective response rate

SECONDARY OUTCOMES:
Disease control rate | Baseline up to approximately 6 months
  t refers to the proportion of patients whose tumor volume control (shrinkage or enlargement) reaches a predetermined value and can maintain the minimum required duration. According to the RECIST criteria (version 1.1), during the treatment period or within 30 days after the discontinuation of the investigational drug, it is the sum of the percentage of subjects who achieve complete response (CR), partial response (PR), and stable disease (SD)
Progression-free survival | Baseline up to approximately 12 months
  It refers to the time from the first administration of the regimen to the first occurrence of disease progression or death due to any cause in the subjects.
Overall survival | Baseline up to approximately 12 months]
  The time from randomization to death due to any cause in the subjects
Duration of response | Baseline up to approximately 12 months
  It refers to the time from the first report of objective tumor partial or complete response (based on the earlier occurrence) to the first occurrence of disease progression or death in the subjects
Clinical benefit rate | Baseline up to approximately 12 months
  The ratio of subjects who achieve complete response (CR) or partial response (PR) or maintain stable disease (SD) .
progression-free survival rate | Baseline up to approximately 12 months
  The percentage of patients who have not experienced disease progression or death due to any cause after receiving the therapy, among the evaluable patients for efficacy.
overall survival rate | Baseline up to approximately 12 months]
  The percentage of patients who died due to any cause after receiving therapy among all enrolled patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital (CAMS&PUMCH), Beijing, Beijing Municipality, China